CLINICAL TRIAL: NCT02300428
Title: Health Economics of the Use of Ferrous Iron Salts in Primary Care in the UK.
Status: Completed | Type: Observational
Sponsor: dora pereira (Other Government)
Collaborators: University of Cambridge (Other); Bangor University (Other); University of Oxford (Other)
Responsible Party: Sponsor-Investigator, dora pereira, Senior Investigator Scientist, Medical Research Council
Organization: Medical Research Council (Other Government)
Other Study IDs: 6531
Record Dates: First submitted 2014-11-24; First posted 2014-11-25 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Anemia
Keywords: iron deficiency
MeSH Terms: conditions — Anemia; Iron Deficiencies | interventions — Iron; ferrous fumarate; ferrous gluconate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1-year cohort: Patients with at least 1 prescription of any oral iron preparation in the last 2 years and who have at least 1 year of follow up data post-prescription.
  It is anticipated that ca. 123,000 patients in CPRD fulfil this criteria.
  Interventions: Dietary Supplement: oral iron
- 10-year cohort: All pre-menopausal women (18-45 years old) with at least 1 prescription of one ferrous iron salt (i.e. sulphate, fumarate and gluconate) since January 2000.
  It is anticipated that ca. 299,000 patients in CPRD fulfil this criteria.
  Interventions: Dietary Supplement: oral iron

INTERVENTIONS:
Dietary Supplement: oral iron — BNF code for section 9.1.1.1 (Oral iron preparations for iron-deficiency anaemias)
  Other Names: Dried ferrous sulphate tablets 200mg; Ferrous fumarate tablets 210mg; Ferrous gluconate tablets 300mg; Ferrous fumarate tablets 322mg (incl. Fersaday); Ferrous fumarate capsules 305mg (incl. Galfer); Dried ferrous sulphate MR tab 325mg (incl. Ferrograd)

SUMMARY:
Iron deficiency anaemia (IDA) affects approximately 4.7 million of people in the UK, with children and pre-menopausal women being at higher risk (1). Each year more than 6.8 million prescriptions for oral iron are filled in England alone (NHS Information Centre data). However, gastrointestinal symptoms limit adherence in 10-30% of otherwise healthy patients (2-4) and in up to 50% of patients with gastrointestinal disorders (5). Simple ferrous iron salts constitute the vast majority of currently prescribed oral iron because these are cheap and well absorbed. However, they are also poorly tolerated and thus, we believe, are expensive to the NHS.

Funded by the Medical Research Council, we have developed an alternative oral iron supplement, that we name IHAT (iron hydroxide adipate tartrate), as an efficacious therapy for IDA with minimal side-effects.

In the study proposed here we aim to assess the total health cost associated with current oral iron supplements and, hence, define the clinical unmet need for alternative treatments. We will use Clinical Practice Research Datalink (CPRD) GOLD data to (i) estimate the pattern of prescribing to oral iron in primary care in the general population and (ii) develop a health economics model in pre-menopausal women. These data will provide evidence for the total health system costs associated with current oral iron treatment. Furthermore, this study will provide data from which the cost-effectiveness and total health system costs of alternative effective and treatments with minimal side-effects could be estimated.

DETAILED DESCRIPTION:
Our research objective is to gather evidence for the unmet clinical need for safe, low-side-effect oral iron in the UK.

To achieve this objective we aim to determine:

1. Pattern of prescribing to oral iron in primary care in GP practices in England: estimate prescription rates, efficacy and intolerance of treatment with all forms of currently prescribed oral iron.
2. Health economics of the use of ferrous iron salts in primary care: estimate patterns of individual response to treatment; determine the costs of ferrous iron (sulphate, fumarate and gluconate) therapy in pre-menopausal women in primary care, and develop a cost-effectiveness model for alternative treatments with minimal side-effects.

ELIGIBILITY:
Inclusion Criteria:

* patients prescribed oral iron in primary care practices included in the UK CPRD database

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For the 1-year cohort study we are not defining a sub-population group and will investigate all individuals (adults and children) prescribed any type of oral iron at least once in the time period assessed, although a breakdown by key sociodemographic (age, gender, ethnicity) will be conducted.
  For the 10-year plus cohort study, pre-menopausal women in receipt of ferrous iron supplements are our study population of interest.
  Pre-menopausal women are the population group with the largest number of individuals affected (nearly 2M) by IDA in the UK, mainly because dietary iron intake does not sufficiently offset menorrhagic iron losses.
Sampling Method: Probability Sample
Enrollment: 406902 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Prescription rate | 12 months
  number of prescriptions of iron supplements issued at the patient level in the year
Health Economics Modelling | 10 years
  In this analysis we will determine the following to parameterise the model that will be based on the cohort study over a 10 years period:
  i) Frequency of repeat oral iron prescriptions, ii) Number of hospital admissions, i) Incidence of gastrointestinal side-effects, ii) Treatment cessation rate iii) Haemoglobin changes
  The basis for the model will be the above data extracted from the CPRD, further informed by publicly available clinical trial data.

SECONDARY OUTCOMES:
Efficacy | 12 months
  increase in Hb of at least 2 g/dL or to >12 g/dL
Gastrointestinal intolerance | 12 months
  At least one event of i. change in product; ii. reduction in dose; iii cessation of treatment with no improvement in Hb during the 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dora Pereira, PhD, Principal Investigator — MRC Human Nutrition Research
Locations (1):
- MRC Human Nutrition Research, Cambridge, Cambridgeshire, United Kingdom